CLINICAL TRIAL: NCT05963126
Title: Modified Urine Fetuin A as a Predictor of Deterioration of Renal Function in Patients With Resistant and Non-resistant Hypertension
Brief Title: Fetuin A as a Predictor of Deterioration of Renal Function in Hypertonic Patients
Status: Recruiting | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: MHUFA-hypertension CKD; RVO-FNOs/2023 17 (Other Grant/Funding Number: University Hospital Ostrava)
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Arterial Hypertension
Keywords: Arterial Hypertension; Resistant Arterial Hypertension; Chronic Kidney Disease; Fetuin A; DNLite IVD103
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples of urine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with hypertension, resistant hypertension, and secondary hypertension: Patients with arterial hypertension, resistant arterial hypertension, and secondary hypertension.
  Interventions: Other: No intervention.

INTERVENTIONS:
Other: No intervention. — No intervention.

SUMMARY:
Commonly used parameters (creatinine, estimated glomerular filtration rate, and urine albumin/creatinine ratio) for prediction of decline of renal function are sensitive for advanced kidney impairment. Modified human urine Fetuin A (urine Fetuin A) with specific modification in urine (Fetuin A) can earlier predict the progression of kidney disease in patients with diabetes. Studies evaluating urine Fetuin A in hypertonic patients are still lacking.

DETAILED DESCRIPTION:
Arterial hypertension and diabetes are the most common cause of chronic kidney disease. Commonly used parameters for the evaluation of renal function (plasma creatinine, estimated glomerular filtration rate, and urine albumin/creatinine ratio) are sensitive to advanced kidney disease. Parameters predicting early kidney impairment are still lacking. Modified human urine Fetuin A with specific modification in urine (urine Fetuin A) presents a new biomarker that seems to be promising in the early prediction of kidney disease in patients with diabetes without microalbuminuria. Studies evaluating urine Fetuin A in hypertonic patients are still lacking.

ELIGIBILITY:
Inclusion Criteria:

* Arterial hypertension treated by at least one antihypertensive agent

Exclusion Criteria:

* Diabetes mellitus of any type, defined as fasting glucose >7,0 mmol/l or any glycemia >11,0 mmol/l, or HbA1c>48 mmol/mol
* Decompensated arterial hypertension defined as office blood pressure >180/110 mmHg or on Ambulatory Blood Pressure Monitoring (ABPM)
* Patient with renal replacement therapy
* Present rheumatoid disease (rheumatoid arthritis, systemic lupus, sclerodermia, dermatomyositis, Inflammatory Bowel Disease, etc.), positivity of antinuclear antibody (ANA) / extractable nuclear antigen (ENA) screening
* Acute infection defined as C-Reactive Protein (CRP) >50 mg/l
* Severe impairment of liver function defined as cirrhosis, Alanine Transaminase or ASpartate Transferase (ALT or AST) >10 µkat/l
* Terminal incurable illness

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hypertension and resistant hypertension followed-up in the Hypertension excellence centre and Lipid centre in University Hospital Ostrava.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Glomerular filtration rate | 1 year
  Decline of glomerular filtration rate in 1-year follow-up of each patient in a total of 3 visits at times: 0 months, 6 months, and 12 months.

SECONDARY OUTCOMES:
Urine biomarker DNLite IVD103 - primary aim | 1 year
  Evaluation of urine biomarker DNLite IVD103 and its ability to predict deterioration of renal function defined as a decline of glomerular filtration rate in patients with arterial hypertension, resistant arterial hypertension, and secondary hypertension. Diabetic nephropathy in vitro diagnostics (DNLite IVD103) is a colorimetric immunoassay intended for quantitative measurement of unique Fetuin-A with specific post-translational modification in human urine.
Urine biomarker DNLite IVD103 - secondary aim | 1 year
  Evaluation of urine biomarker DNLite IVD103 and its ability to predict deterioration of renal function defined in patients with manifested cardiovascular disease, dyslipidemia (yes/no).
Urine biomarker DNLite IVD103 - correlation | 1 year
  Evaluation of the correlation of biomarker DNLite IVD103 in patients' plasma and in urine (yes/no).

CONTACTS AND LOCATIONS:
Overall Officials: Zdeněk Ramík, MD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, - Department of Internal Medicine and Cardiology, Ostrava, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data with other researchers.

REFERENCES:
- See also: The DNlite Test - Products - BIOPREVENTIVE MEDICINE — https://bpmbiotech.com